CLINICAL TRIAL: NCT05226949
Title: Host RNA Expression Profiles and Protein Biomarkers in Neonatal Herpes Simplex Virus Infection
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Statens Serum Institut (Other)
Responsible Party: Principal Investigator, Kia Hee Schultz Dungu, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: H-21009288-HSV
Record Dates: First submitted 2022-01-27; First posted 2022-02-07 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Neonatal Herpes Simplex Infection; Neonatal HSV Infection; Neonatal Infection; Newborn; Infection; Herpes Simplex Virus Infection; Neonatal Sepsis; Neonatal Death; Viral Infection
MeSH Terms: conditions — Neonatal herpes; Infections; Herpes Simplex; Neonatal Sepsis; Perinatal Death; Virus Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Dried blood spot samples will be obtained from the Danish Neonatal Screening Biobank, Statens Serum Institut. RNA sequencing and proteomic analyses (in total 12 ul whole blood) will be performed at the Danish Center for Neonatal Screening, Department of Congenital Disorders, Statens Serum Institut.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: 54 newborns with neonatal HSV infection.
  Interventions:
  Diagnostic test and disease pathogenesis: Host RNA expression profiling by RNA sequencing and proteomic analyses. Cases will be randomly assigned to a "Discovery Cohort" (identification of diagnostic RNA and proteomic profiles).
- Controls: 108 newborns without infection.
  Interventions:
  Diagnostic test and disease pathogenesis: Host RNA expression profiling by RNA sequencing and proteomic analyses. Controls will be randomly assigned to a "Discovery Cohort" (identification of diagnostic RNA and proteomic profiles).

SUMMARY:
This study seeks to identify and test host RNA expression profiles in context to protein biomarkers in dried blood spot samples as novel diagnostic markers of neonatal herpes simplex virus infection and to improve the understanding of the pathogenesis of the disease.

DETAILED DESCRIPTION:
Background:

Herpes Simplex Virus (HSV) infection in newborns is uncommon but can be devastating and is associated with significant morbidity and mortality. The diagnosis of neonatal HSV infection is challenging because maternal genital herpes often is asymptomatic and the clinical presentation in newborns can be nonspecific, especially in the early disease stages. This results in late diagnosis and potentially terrible consequences for the newborn. The reason why some newborns develop severe disease due to HSV infection is unknown. It has been suggested that immunologic differences in early infancy are the key to further advances. Host RNA expression profiling, transcriptomics, of the host response to infections has shown great potential as clinical tool for diagnostics and for unveiling molecular disease mechanisms. As previously shown, reliable host RNA expression data can be obtained from neonatal dried blood spot (DBS) samples by RNA-sequencing. Proteomic analysis has the potential to simultaneously identify hundreds of protein biomarkers and immune cell populations allowing for detailed mapping of disease immunological pathways.

Method:

A nationwide retrospective case-control study of all newborns with HSV infection in Denmark from 2010 through 2019. DBS samples will be obtained from the Danish Neonatal Screening Biobank, Statens Serum Institut. RNA sequencing and proteomic analyses will be performed at the Danish Center for Neonatal Screening, Department of Congenital Disorders, Statens Serum Institut. Cases will be randomly assigned to a "Discovery cohort" and compared to a control group of newborns matched on gestational age, sex and birthweight will be included.

Time frame:

Sample identification/recruiting: January 1st to January 31st 2022. Sample analysis (RNA sequencing and proteomic analysis): February 1st to April 30th 2022.

Perspectives:

New molecular-based diagnostic tools complementary to conventional methods may improve early diagnosis of neonatal HSV infections and lead to optimised management. In addition, understanding of the pathogenesis at a molecular level of severe disease manifestations of the disease, could form the basis for development of novel interventions for better prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. cases of newborns aged 0-28 days with verified HSV infection (positive HSV PCR in blood, cerebrospinal fluid and/or swab sample)
2. controls of newborns without infection matched on gestational age, sex and birthweight

Exclusion Criteria:

1. dried blood spot samples that are not allowed to be used for research
2. dried blood spots samples containing insufficient amount of blood for research

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns aged 0-28 days with verified HSV infection in Denmark from 2010 through 2019.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Host RNA expression and proteomic profiles | Admission, age 0-28 days
  To identify specific host RNA expression and proteomic profiles in dried blood spot samples from newborns with HSV infection

SECONDARY OUTCOMES:
Disease pathogenesis | Admission, age 0-28 days
  Mapping of disease immunological pathways by simultaneous host RNA expression profiling and proteomic analysis
Application of known host RNA profiles | Admission, age 0-28 days
  To test host RNA profiles published in other studies, e.g. based on the genes IFI44L and FAM89A

CONTACTS AND LOCATIONS:
Overall Officials: Kia Hee Schultz Dungu, MD, Principal Investigator — Rigshospitalet, Denmark; Ulrikka Nygaard, Ass Prof PhD, Study Chair — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Department of Paediatrics and Adolescent Medicine, Rigshospitalet, Copenhagen
  - Department of Congenital Disorders, Statens Serum Institut, Copenhagen

IPD SHARING:
Plan to Share IPD: Undecided